CLINICAL TRIAL: NCT02816918
Title: Extraluminal Use of the Bronchial Blocker of Univent Tube During Adult One-lung Ventilation
Brief Title: Extraluminal Use of the Bronchial Blocker of Univent Tube
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 995866
Record Dates: First submitted 2016-06-09; First posted 2016-06-29 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-08

CONDITIONS: Therapeutic Procedural Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extraluminal use of Univent Blocker (Experimental): Patients assigned to the Extraluminal use of Univent Blocker group were first inserted Univent bronchial Blocker into the glottis via direct laryngoscopy then advanced the Blocker to the target bronchus until slight resistance was encountered.A conventional tracheal tube with appropriate size was intubated via direct laryngoscopy into the appropriate depth, inflating the tracheal tube cuff, and fixing the tube firmly at the patient's mouth with cloth tape .
  So the Univent Blocker Extraluminal of the endotracheal tube,then the fibreoptic bronchoscopy was inserted into the tracheal tube and guided bronchial blocker cuff to the target main bronchus under direct vision
  Interventions: Device: Extraluminal use of Univent bronchial Blocker
- Innerluminal use of Univent Blocker (Experimental): Patients in Innerluminal use of Univent Blocker group: When the endotracheal tube had been intubated via direct laryngoscopy, the bronchial blocker was advanced Innerluminal of the endotracheal tube and directed into the right or left mainstem bronchus, then the fibreoptic bronchoscopy was inserted into the tracheal tube. After further pushing and twisting, the bronchial blocker tube will move into the mainstem bronchus under direct vision by FOB.the tracheal tube cuff is inflated with the tube being fixed firmly at the patient's mouth with cloth tape
  Interventions: Device: Innerluminal use Univent bronchial Blocker

INTERVENTIONS:
Device: Extraluminal use of Univent bronchial Blocker — Patients assigned to the Extraluminal use of Univent Blocker group were first inserted Univent bronchial Blocker into the glottis via direct laryngoscopy then advanced the Blocker to the target bronchus until slight resistance was encountered.A conventional tracheal tube with appropriate size was intubated via direct laryngoscopy into the appropriate depth, inflating the tracheal tube cuff, and fixing the tube firmly at the patient's mouth with cloth tape .
  So the Univent Blocker Extraluminal of the endotracheal tube,then the fibreoptic bronchoscopy was inserted into the tracheal tube and guided bronchial blocker cuff to the target main bronchus under direct vision
  Arms: Extraluminal use of Univent Blocker
Device: Innerluminal use Univent bronchial Blocker — Patients in Innerluminal use of Univent Blocker group: When the endotracheal tube had been intubated via direct laryngoscopy, the bronchial blocker was advanced Innerluminal of the endotracheal tube and directed into the right or left mainstem bronchus, then the fibreoptic bronchoscopy was inserted into the tracheal tube. After further pushing and twisting, the bronchial blocker tube will move into the mainstem bronchus under direct vision by FOB.the tracheal tube cuff is inflated with the tube being fixed firmly at the patient's mouth with cloth tape
  Arms: Innerluminal use of Univent Blocker

SUMMARY:
intends to evaluate the feasibility and security issues of univent bronchial blockers outside the single lumen endotracheal tube for one- lung ventilation in left thoracic surgery patients.

DETAILED DESCRIPTION:
One-lung ventilation is desirable for Several clinical procedures, such as thoracic,pulmonary, and cardiac surgery to facilitate lung exposure for these surgical procedures by collapsing the lung and most commonly used device is the double-lumen tube (DLT) for this surgical procedures.Bronchial blockers (BBs), such as univent tube with an bronchial Blocker, has more advantages than the double-lumen tube: no need exchange tube when mechanical ventilation is required postoperative, easier insertion,less postoperative sore throat (ST) and hoarseness. However, BBs requires more time for placement and more difficult to position, especially patients undergoing left-side thoracic surgery. So, this study intends to evaluate the feasibility and security issues of univent bronchial blockers outside the single lumen endotracheal tube for one- lung ventilation in left thoracic surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* sixty patients undergoing left thoracic surgery
* ASA classifications of I-II, modified Mallampati classification of 1 or 2, requiring general anesthesia were included.

Exclusion Criteria:

* age younger than 18 yr or older than 70 yr
* BMI>30 kg/m2
* with upper respiratory tract infection,asthma
* Abnormalities of the heart, brain, liver, lung, kidney and coagulation functions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
time for positioning | 15 min

SECONDARY OUTCOMES:
frequency of malpositions | 5 min
frequency of fiberoptic | 10 min

CONTACTS AND LOCATIONS:
Overall Officials: Ximing Qi, Study Director — The First Hospital of Qinhuangdao
Locations (1):
- 中国, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes